CLINICAL TRIAL: NCT00629902
Title: Impact of Prosthesis-Patient Mismatch on Clinical Outcomes After Mitral Valve Replacement
Brief Title: Heart Valve Prosthesis-Patient Mismatch
Status: Completed | Type: Observational
Sponsor: Florence Nightingale Hospital, Istanbul (Other)
Responsible Party: Saide Aytekin, Florence Nightingale Hospital
Other Study IDs: AT-1974
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Heart Valve Diseases
Keywords: Heart valve prosthesis
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A1: Patients with prosthesis-patient mismatch after mitral valve replacement
- A2: Patients without prosthesis mismatch after mitral valve replacement

SUMMARY:
The purpose of this study is to determine the frequency of prosthesis-patient mismatch after mitral valve replacement and its effect on clinical outcomes.

DETAILED DESCRIPTION:
Mitral valve replacement (MVR) is associated with higher short and long term mortality than aortic valve replacement or mitral valve repair. The suboptimal results of MVR underline the importance of identifying and preventing prosthesis- patient mismatch. The effective orifice area (EOA) of prosthetic valves used for MVR is often too small in relation to body size, thus causing a mismatch between valve EOA and transvalvular flow. As a consequence, normally functioning mitral prostheses often have relatively high gradients that are similar to those found in patients with mild to moderate mitral stenosis. Residual pressure gradients across mitral prostheses delay the regression of left atrial and pulmonary arterial hypertension. Pulmonary hypertension may cause rightsided failure and is an important risk factor for morbidity and mortality in patients with cardiovascular diseases. However data about the frequency of prosthesis-patient mismatch after mitral valve replacement and its effect on clinical outcome is inconclusive. Predetermined outcomes will be evaluated in the clinical course of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years with a clinical condition of mitral valve prosthesis

Exclusion Criteria:

* Evidence of prosthesis valve dysfunction (dehisence, endocarditis or thrombus of prosthetic mitral valve)
* Concomitant aortic valve prosthesis and tricuspid valve prosthesis
* Presence of > +2 aortic valve regurgitation and/or mild aortic stenosis
* Prosthetic mitral valve replacement operation < 6 months
* Left ventricular ejection fraction < 50%
* Chronic obstructive pulmonary disease
* Concomitant hypertrophic cardiomyopathy, atrial septal defect
* Patients with poor ehocardiographic window

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saide Aytekin, Professor, Principal Investigator — T.C. Istanbul Bilim University, Medical Faculty, Florence Nightingale Hospital, Division of Cardiology
Locations (1):
- T.C. Bilim University, Medical Faculty, Florence Nightingale Hospital, Division of Cardiology, Istanbul, Sisli, Turkey (Türkiye)

REFERENCES:
- [Background] Totaro P, Argano V. Patient-prosthesis mismatch after mitral valve replacement: myth or reality? J Thorac Cardiovasc Surg. 2007 Sep;134(3):697-701. doi: 10.1016/j.jtcvs.2007.04.031. PMID 17723820
- [Background] Li M, Dumesnil JG, Mathieu P, Pibarot P. Impact of valve prosthesis-patient mismatch on pulmonary arterial pressure after mitral valve replacement. J Am Coll Cardiol. 2005 Apr 5;45(7):1034-40. doi: 10.1016/j.jacc.2004.10.073. PMID 15808760
- [Background] Magne J, Mathieu P, Dumesnil JG, Tanne D, Dagenais F, Doyle D, Pibarot P. Impact of prosthesis-patient mismatch on survival after mitral valve replacement. Circulation. 2007 Mar 20;115(11):1417-25. doi: 10.1161/CIRCULATIONAHA.106.631549. Epub 2007 Mar 5. PMID 17339554